CLINICAL TRIAL: NCT06072976
Title: The Influence of Feeding Source on the Gut Microbiome and Time to Full Feeds in Neonates With Congenital Gastrointestinal Pathologies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Katie, Katie Strobel, MD, Seattle Children's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00004330: CGP Milk
Record Dates: First submitted 2023-08-08; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Gastrointestinal Complication; Intestinal Obstruction; Gastroschisis; Hirschsprung Disease; Omphalocele; Midgut Volvulus
MeSH Terms: conditions — Intestinal Obstruction; Gastroschisis; Hirschsprung Disease; Hernia, Umbilical; Volvulus Of Midgut | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exclusive human milk (Experimental): Mothers will consent to providing DHM if MOM is not available. If the infant reaches 100 ml/kg/day of feeds (one feed advancement prior to full feeds) and MOM remains unavailable, they will transition to formula in preparation for discharge. Infants cannot be discharged on donor milk.
  Interventions: Dietary Supplement: Exclusive Human Milk
- Standard of care (Experimental): Mothers will consent to providing DHM (if qualifies per hospital policy) or formula if MOM is not available. Infants are only eligible to receive donor milk only if 1) MOM is not available 2) if infant initiates feeds before day 3 of age. The donor milk feed would be stopped on day 5 of age. After day five of age, the infant will receive formula if MOM is not available. This is congruent with the current donor milk policy (see Policy #12785). It is highly unlikely given these infants would receive any donor milk because these infants require surgery and often are waiting return of bowel function . The median age of initiation of feeds is 12 days of age for infants with gastroschisis (PMID: 33647253) which exceeds the days of what the hospital policy says for eligibility which is initiates feed before day 3 of age. If the infant does not qualify for any donor milk and MOM is not available, the infant will receive formula
  Interventions: Dietary Supplement: Standard of Care

INTERVENTIONS:
Dietary Supplement: Standard of Care — Standard of care arm: Mothers will consent to providing DHM (if qualifies per hospital policy) or formula if MOM is not available. Infants are only eligible to receive donor milk only if 1) MOM is not available 2) if infant initiates feeds before day 3 of age. The donor milk feed would be stopped on day 5 of age.
  Arms: Standard of care
Dietary Supplement: Exclusive Human Milk — Mothers will consent to providing DHM if MOM is not available. If the infant reaches 100 ml/kg/day of feeds (one feed advancement prior to full feeds) and MOM remains unavailable, they will transition to formula in preparation for discharge. Infants cannot be discharged on donor milk.
  Arms: Exclusive human milk

SUMMARY:
This study explores the use of an exclusive human milk diet versus standard feeding practices to compare the influence on feeding outcomes and the gut bacteria in infants with intestinal differences.

ELIGIBILITY:
Inclusion Criteria:

* Infants with gastroschisis, giant omphalocele, intestinal atresia, mid-gut volvulus, hirschsprungs disease.

Exclusion Criteria:

1. Infant has already been on feeds
2. Infants <34 weeks gestation
3. Parents with contraindications to providing milk (i.e. drug use-cocaine, fentanyl, meth BUT oxy/suboxone/marijuana OK)
4. Complicated gastroschisis
5. Short gut syndrome
6. Additional congenital anomalies that affect ability to tolerate milk (i.e. cyanotic congenital heart disease BUT kidney disease ok)

Ages: 0 Days to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2025-06-09 (Estimated); Study Completion 2025-06-09 (Estimated)

PRIMARY OUTCOMES:
Time to full feed | From birth to 120 days or until discharge
  : In infants with congenital gastrointestinal pathologies (gastroschisis, giant omphalocele, atresia, midgut volvulus, Hirschsprung disease, CGP), to determine if use of an exclusive human milk diet will decrease the number of days to full feeding volume (120 ml/kg/day) (29 subjects per power calculation) compared to human milk/formula

SECONDARY OUTCOMES:
Central line infection rate | up to 120 days or discharge
  To compare rate of central line infections in infants given exclusive human milk versus infants given standard care.
Portion of parents own milk at time of discharge | Up to 120 days or discharge
  : To compare proportion of parents providing any/exclusive mother's own milk (MOM) at discharge in infants given exclusive human milk arm versus standard care arm
Gut Microbiome Relative Abundance and Diversity | Up to 120 days or discharge
  To examine if utilization of donor milk when mother's own milk is insufficient alters the infant's gut microbiome alpha diversity and beta diversity and bacterial relative abundances
Mother's milk microbiome relative abundance and diversity | Up to 120 days or discharge
  To discern how mother's own milk microbiome differs from donor milk microbiome relative abundances and diversity. We will examine how the milk microbiomes influences the infant's gut microbiome and time to full feeds.
Concentrations of Antigen-specific immunoglobulins | From birth to 120 days or discharge
  To compare total and antigen-specific immunoglobulins in donor milk versus MOM

CONTACTS AND LOCATIONS:
Overall Officials: Katie Strobel, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

REFERENCES:
- [Background] Varma S, Bartlett EL, Nam L, Shores DR. Use of Breast Milk and Other Feeding Practices Following Gastrointestinal Surgery in Infants. J Pediatr Gastroenterol Nutr. 2019 Feb;68(2):264-271. doi: 10.1097/MPG.0000000000002128. PMID 30119100
- [Background] Hoban R, Khatri S, Patel A, Unger SL. Supplementation of Mother's Own Milk with Donor Milk in Infants with Gastroschisis or Intestinal Atresia: A Retrospective Study. Nutrients. 2020 Feb 24;12(2):589. doi: 10.3390/nu12020589. PMID 32102333
- [Background] Bergner EM, Shypailo R, Visuthranukul C, Hagan J, O'Donnell AR, Hawthorne KM, Abrams SA, Hair AB. Growth, Body Composition, and Neurodevelopmental Outcomes at 2 Years Among Preterm Infants Fed an Exclusive Human Milk Diet in the Neonatal Intensive Care Unit: A Pilot Study. Breastfeed Med. 2020 May;15(5):304-311. doi: 10.1089/bfm.2019.0210. Epub 2020 Apr 16. PMID 32298596
- [Background] Hair AB, Rechtman DJ, Lee ML, Niklas V. Beyond Necrotizing Enterocolitis: Other Clinical Advantages of an Exclusive Human Milk Diet. Breastfeed Med. 2018 Jul/Aug;13(6):408-411. doi: 10.1089/bfm.2017.0192. Epub 2018 Jun 7. PMID 29877722
- [Background] Murthy S, Parker PR, Gross SJ. Low rate of necrotizing enterocolitis in extremely low birth weight infants using a hospital-based preterm milk bank. J Perinatol. 2019 Jan;39(1):108-114. doi: 10.1038/s41372-018-0235-3. Epub 2018 Oct 5. PMID 30291318
- [Background] Fleig L, Hagan J, Lee ML, Abrams SA, Hawthorne KM, Hair AB. Growth outcomes of small for gestational age preterm infants before and after implementation of an exclusive human milk-based diet. J Perinatol. 2021 Aug;41(8):1859-1864. doi: 10.1038/s41372-021-01082-x. Epub 2021 May 19. PMID 34012050
- [Background] Hair AB, Good M. Dilemmas in feeding infants with intestinal failure: a neonatologist's perspective. J Perinatol. 2023 Jan;43(1):114-119. doi: 10.1038/s41372-022-01504-4. Epub 2022 Sep 20. PMID 36127395
- [Background] Strobel KM, Kramer K, Rottkamp CA, Uy C, Moyer L, Fernandez E, Elashoff D, Sabnis A, and Calkins KL. Implementation of a Nutritional Pathway Across California Hospitals Improves Linear Growth in Neonates with Gastroschisis: A University of California Fetal Consortium Study. Pediatric Academic Societies, 4/22/2022, Denver, CO.
- [Background] Hodgson EC, Livingston MH, Robinson T, Farrokhyar F, Walton JM. Use of breast milk in infants with uncomplicated gastroschisis: A retrospective cohort study. J Pediatr Surg. 2022 May;57(5):840-845. doi: 10.1016/j.jpedsurg.2021.12.045. Epub 2022 Jan 13. PMID 35058060
- [Background] Spatz DL, Robinson AC, Froh EB. Cost and Use of Pasteurized Donor Human Milk at a Children's Hospital. J Obstet Gynecol Neonatal Nurs. 2018 Jul;47(4):583-588. doi: 10.1016/j.jogn.2017.11.004. Epub 2017 Dec 6. PMID 29221672
- [Background] Kumbhare SV, Jones WD, Fast S, Bonner C, Jong G', Van Domselaar G, Graham M, Narvey M, Azad MB. Source of human milk (mother or donor) is more important than fortifier type (human or bovine) in shaping the preterm infant microbiome. Cell Rep Med. 2022 Sep 20;3(9):100712. doi: 10.1016/j.xcrm.2022.100712. Epub 2022 Aug 26. PMID 36029771
- [Background] Demers-Mathieu V, Huston RK, Markell AM, McCulley EA, Martin RL, Spooner M, Dallas DC. Differences in Maternal Immunoglobulins within Mother's Own Breast Milk and Donor Breast Milk and across Digestion in Preterm Infants. Nutrients. 2019 Apr 24;11(4):920. doi: 10.3390/nu11040920. PMID 31022910